CLINICAL TRIAL: NCT02058134
Title: CardioPAT Project - Reducing the Need for Allogenic Blood Transfusion After On-pump Cardiac Surgery With Intra- and Postoperative Use of a New Device: a Randomized Trial
Brief Title: The CardioPAT Project: A Randomized Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to other trials in the department
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Erika Nodin, Research Scholar, Rigshospitalet, Denmark
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-3-2013-169
Record Dates: First submitted 2014-02-06; First posted 2014-02-07 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2016-08

CONDITIONS: Coronary Artery Disease; Aortic Stenosis; Aortic Insufficiency; Mitral Insufficiency; Aortic Aneurysm
MeSH Terms: conditions — Coronary Artery Disease; Aortic Valve Stenosis; Aortic Valve Insufficiency; Mitral Valve Insufficiency; Aortic Aneurysm

ARMS (2):
- Control group (No Intervention)
- Interventional group (Experimental): For patients in the interventional group we use a CardioPAT cell saver intra- and postoperatively.
  Interventions: Device: cardioPAT cell saver

INTERVENTIONS:
Device: cardioPAT cell saver
  Arms: Interventional group

SUMMARY:
The purpose of this study is to determine whether intra- and postoperative use of the cardioPAT® cell saver decreases the need for allogenic red blood cell transfusion in patients, who undergo open heart surgery (with cardiopulmonary bypass) and preoperatively have an increased risk for bleeding.

DETAILED DESCRIPTION:
This scientific study will be conducted as a randomized controlled trial with N = 146, and therefore n = 2 x 73.

Randomization will be carried out as a simple 1:1 randomization in to the following groups:

1. Control group: undergo heart surgery with blood conserving strategies that are currently standard routine at Rigshospitalet.
2. Interventional group: undergo heart surgery with intra- and postoperative use of the cardioPAT cell saver. The cardioPAT collects blood from the operative site and from the chest tubes, thereafter it washes and concentrates the red blood cells. This blood can then be returned to the patient. Furthermore, this group will also receive the same blood conserving strategies as the control group.

Randomization will be stratified for the inclusion criteria to ensure that the two groups have the same amount of women, men with a hemoglobin under 8 mmol/l and men over 75 years with double procedures.

All legally competent adults who receive an on-pump open heart surgery at the Department of Cardiothoracic Surgery at Rigshospitalet will be screened for participation in this trial.

Inclusion criteria:

Patients with an increased risk for bleeding, who undergo open heart surgery, that is:

* Women
* Men with a hemoglobin < 8mmol/L
* Men > 75 years of age with combined procedures, that is f.ex. combined CABG and valve surgery, regardless of preoperative hemoglobin level

Exclusion criteria:

* Re-operation within the first 24 hours
* Known clotting disorders (coagulopathy) or hematological diseases
* Sepsis, f ex due to Endocarditis
* Patients who are already enrolled in other studies, where data from the studies are at risk of interfering with each other
* Jehovah's witnesses
* Acute surgery (< 24 hours)

The aim of the study is to investigate:

* Whether the requirement for allogenic transfusion of red blood cells (SAG-M), platelets and fresh frozen plasma to patients, with an increased bleeding risk who undergo open heart surgery, can be decreased with intra- and postoperative use of the cardioPAT® cell saver
* Whether the percentage of patients receiving no transfusion (0 units) is increased with the use of a cardioPAT® cell saver
* The cost-effectiveness of using the cardioPAT® cell saver compared with the current standard treatment
* Hemoglobin and platelet count for the interventional group pre- and postoperatively, as well as at discharge and compare these with the control group
* The composition and quality of the cardioPAT® red blood cell product
* The composition of the cardioPAT® waste product
* The length of stay in the ICU and total hospitalization after cardiac surgery
* The impact on different aspects of coagulation
* The extent of renal impairment in the postoperative period
* The inflammatory response in the postoperative period
* Endothelial injury in in the postoperative period

Sample size calculation:

The standard deviation, for blood transfusion to patients at the Department of Cardiothoracic Surgery, Rigshospitalet, was calculated to ±0,32.

From a clinical point of view a relevant reduction, which would justify a routine use of the CardioPAT® device, would be somewhere between 15-20%. This reduction would result in the Department saving every 1/7 to 1/5 unit of blood. Therefore a difference of 15% will be used for the power calculation.

Sample size was calculated by means of a "Sample Size Calculator" found online at: http://hedwig.mgh.harvard.edu/sample_size/size.html.This power analysis calculated that a total of 146 patients will need to enter this two-treatment parallel-design study. The probability (power) is 80% that the study will detect a treatment difference at a two-sided 0,05 significance level, based on the assumption that the standard deviation of the response variable is 0,32 and the true difference between treatments is set to 0,15 units (15%).

An interim analysis will be conducted after the inclusion of approximately 80 patients. If the results are relevant at this time, the study will stop inclusion here and present the results.

ELIGIBILITY:
Inclusion Criteria:

* All the women
* Men with a hemoglobin < 8mmol/L
* Men > 75 years of age with combined procedures, that is combined CABG and valve surgery, regardless of preoperative hemoglobin level
* Sub-acute patients can be included

Exclusion Criteria:

* Re-operation within the first 24 hours
* Known clotting disorders (coagulopathy) or hematological diseases
* Sepsis, f ex due to Endocarditis
* Patients who are already enrolled in other studies, where data from the studies are at risk of interfering with each other
* Jehovah's witnesses
* Acute surgery (< 24 hours)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2013-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
The rate of allogenic transfusion with red blood cells (SAG-M) | The entire stay at the Department of Cardiothoracic Surgery, Rigshospitalet (approximately one week after surgery)

CONTACTS AND LOCATIONS:
Overall Officials: Erika Nodin, MD, Principal Investigator — Department of Cardiothoracic Surgery, Rigshospitalet, Denmark
Locations (1):
- Department of Cardiothoracic Surgery, Rigshospitalet, Copenhagen, København Ø, Denmark